CLINICAL TRIAL: NCT05123625
Title: A Phase III Randomized Non-inferiority Multicenter Study of PLND Omission in Clinical NMIBC Undergoing Radical Cystectomy
Brief Title: Prognostic Effect of Whether Doing PLND During RC for High-risk NMIBC
Acronym: PLND-Less
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: The Second Affiliated Hospital of Kunming Medical University (Other); Tianjin Medical University Second Hospital (Other); RenJi Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-SR-291.A1
Record Dates: First submitted 2021-09-08; First posted 2021-11-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-05

CONDITIONS: Bladder Cancer
Keywords: High-risk; Lymphadenectomy; Non-muscular invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RC combined with lymph node dissection (No Intervention): When radical cystectomy was performed, pelvic lymph node dissection was also performed.
- Only RC (Experimental): In the intervention group, investigators used a reductive approach. That is, for radical cystectomy, investigators did not perform pelvic lymph node dissection.
  Interventions: Procedure: Reduce surgical procedures

INTERVENTIONS:
Procedure: Reduce surgical procedures — In the intervention group, investigators used a reductive approach. That is, for radical cystectomy, investigators did not perform pelvic lymph node dissection.
  Arms: Only RC

SUMMARY:
There is no consensus on the need for lymph node dissection in radical cystectomy (RC) for high-risk non-muscular invasive bladder cancer (NMIBC). Investigators divided participants at high risk of NMIBC without enlarged lymph nodes as indicated by pelvic MRI into two groups 1:1. One group of participants underwent RC combined with lymph node dissection and the other group of participants only underwent RC. The incidence of complications and PFS/OS at 1, 3, and 5 years were compared.

DETAILED DESCRIPTION:
Bladder cancer is highly prevalent worldwide and approximately 75% of these are non-muscle invasive bladder cancer (NMIBC). For high-risk NMIBC, postoperative intravesical chemotherapy combined with full-dose BCG for 3 years is recommended. Radical cystectomy (RC) is also one of the treatment options, and is recommended for patients with BCG-naïve, BCG-refractory, and recurrent high-grade or carcinoma-in-situ (CIS) bladder cancer after BCG perfusion.

RC combined with pelvic lymph node dissection is the standard treatment for MIBC. Currently, there is no conclusion on the radical treatment of NMIBC, most of NMIBC patients refer to MIBC and also perform pelvic lymph node dissection. However, long operation time, high incidence of lymphatic cyst, lymphatic leakage and other complications, and long recovery time, increase the psychological and economic burden. At present, many studies have showed that the positive rate of lymph nodes in NMIBC patients is low. Investigators also analyzed the data of patients who underwent RC in investigators' center from 2013 to 2019, and found that the positive rate of lymph nodes in 163 NMIBC patients was only 3.07%.

MRI can effectively predict pelvic metastatic lymph nodes, and its sensitivity and negative predictive values have been reported as high as 76.4% and 71.4%. VI-RADS score can effectively judge the muscularity of bladder tumor. Therefore, Investigators proposed whether it is necessary to perform pelvic lymph node dissection in NMIBC patients without enlarged lymph nodes indicated by pelvic MRI. Investigators intended to divide participants at high risk of NMIBC without enlarged lymph nodes as indicated by pelvic MRI into two groups 1:1. One group underwent RC combined with lymph node dissection and the other group only underwent RC. The incidence of complications and PFS/OS at 1, 3, and 5 years were compared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who did not undergo diagnostic transurethral resection of bladder tumor (TURBT): biopsy suggestive of G3/high grade or with CIS or cystoscopic findings of multiple, tumor diameter greater than 3 cm; and VI-RADS score of 1 or 2; and no enlarged lymph nodes detected by MRI.
2. Patients undergoing diagnostic TURBT: pathologically confirmed high-risk NMIBC, a) stage T1; b) G3 or high-grade; c) CIS; d) multiple, recurrent TaG1G2/low-grade bladder cancer patients with >3 cm in diameter. And no enlarged lymph nodes detected on MRI.
3. Benefit from radical cystectomy as assessed by the investigator.
4. Meeting the indications for the procedure: a) absolute neutrophil count ≥ 1.5 *109/L; b) platelets ≥ 100 *109/L; c) hemoglobin ≥ 90 g/L; d) international normalized ratio or activated partial thromboplastin time ≤ 1.5 upper limit of normal (ULN); e) calculated creatinine clearance ≥ 1 ml/s f) serum total bilirubin ≤ 1.5 * ULN; g) AST, ALT and alkaline phosphatase ≤ 2.5 * ULN; h) cardiopulmonary function suggestive of tolerance to major abdominal surgery.
5. No previous history of tumor, lymph node dissection, or immune system-related disease.
6. Age 18 to 75 years.
7. No neoadjuvant therapy.
8. ECOG physical status 0 or 1.
9. Voluntary participation in this trial, ability to provide written informed consent, and understanding and agreement to comply with the requirements of this study and the evaluation schedule.

Exclusion Criteria:

1. Patients with bladder cancer ≥ T2N0M0 confirmed by pathology or assessed by imaging, or with pelvic lymph node enlargement indicated by MRI;
2. The investigator assessed patients who could not tolerate radical cystectomy;
3. Previous systemic chemotherapy or immunotherapy;
4. The presence of active autoimmune diseases requiring systemic treatment or other diseases requiring long-term use of large amounts of hormones and other immunosuppressants;
5. Had undergone major surgery or major trauma within 28 days before enrollment;
6. Received live vaccine within 28 days before enrollment;
7. Severe chronic or active infections requiring systemic antibacterial, antifungal or antiviral therapy within 14 days prior to enrollment;
8. Received any Chinese herbal medicine or proprietary Chinese medicine for cancer control within 14 days before enrollment;
9. Participating in other clinical studies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 5 years after surgery
  progression-free survival

SECONDARY OUTCOMES:
OS | 5 years after surgery
  Overall Survival

OTHER OUTCOMES:
Complication rate | through study completion, an average of 1 year
  Complication rate after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Lu, PhD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burger M, Catto JW, Dalbagni G, Grossman HB, Herr H, Karakiewicz P, Kassouf W, Kiemeney LA, La Vecchia C, Shariat S, Lotan Y. Epidemiology and risk factors of urothelial bladder cancer. Eur Urol. 2013 Feb;63(2):234-41. doi: 10.1016/j.eururo.2012.07.033. Epub 2012 Jul 25. PMID 22877502
- [Background] Babjuk M, Burger M, Comperat EM, Gontero P, Mostafid AH, Palou J, van Rhijn BWG, Roupret M, Shariat SF, Sylvester R, Zigeuner R, Capoun O, Cohen D, Escrig JLD, Hernandez V, Peyronnet B, Seisen T, Soukup V. European Association of Urology Guidelines on Non-muscle-invasive Bladder Cancer (TaT1 and Carcinoma In Situ) - 2019 Update. Eur Urol. 2019 Nov;76(5):639-657. doi: 10.1016/j.eururo.2019.08.016. Epub 2019 Aug 20. PMID 31443960
- [Background] Chang SS, Boorjian SA, Chou R, Clark PE, Daneshmand S, Konety BR, Pruthi R, Quale DZ, Ritch CR, Seigne JD, Skinner EC, Smith ND, McKiernan JM. Diagnosis and Treatment of Non-Muscle Invasive Bladder Cancer: AUA/SUO Guideline. J Urol. 2016 Oct;196(4):1021-9. doi: 10.1016/j.juro.2016.06.049. Epub 2016 Jun 16. PMID 27317986
- [Background] Raj GV, Herr H, Serio AM, Donat SM, Bochner BH, Vickers AJ, Dalbagni G. Treatment paradigm shift may improve survival of patients with high risk superficial bladder cancer. J Urol. 2007 Apr;177(4):1283-6; discussion 1286. doi: 10.1016/j.juro.2006.11.090. PMID 17382713
- [Background] Witjes JA, Bruins HM, Cathomas R, Comperat EM, Cowan NC, Gakis G, Hernandez V, Linares Espinos E, Lorch A, Neuzillet Y, Rouanne M, Thalmann GN, Veskimae E, Ribal MJ, van der Heijden AG. European Association of Urology Guidelines on Muscle-invasive and Metastatic Bladder Cancer: Summary of the 2020 Guidelines. Eur Urol. 2021 Jan;79(1):82-104. doi: 10.1016/j.eururo.2020.03.055. Epub 2020 Apr 29. PMID 32360052
- [Background] Chang SS, Bochner BH, Chou R, Dreicer R, Kamat AM, Lerner SP, Lotan Y, Meeks JJ, Michalski JM, Morgan TM, Quale DZ, Rosenberg JE, Zietman AL, Holzbeierlein JM. Treatment of Non-Metastatic Muscle-Invasive Bladder Cancer: AUA/ASCO/ASTRO/SUO Guideline. J Urol. 2017 Sep;198(3):552-559. doi: 10.1016/j.juro.2017.04.086. Epub 2017 Apr 26. PMID 28456635
- [Background] Bruins HM, Huang GJ, Cai J, Skinner DG, Stein JP, Penson DF. Clinical outcomes and recurrence predictors of lymph node positive urothelial cancer after cystectomy. J Urol. 2009 Nov;182(5):2182-7. doi: 10.1016/j.juro.2009.07.017. Epub 2009 Sep 15. PMID 19758623
- [Background] Karl A, Carroll PR, Gschwend JE, Knuchel R, Montorsi F, Stief CG, Studer UE. The impact of lymphadenectomy and lymph node metastasis on the outcomes of radical cystectomy for bladder cancer. Eur Urol. 2009 Apr;55(4):826-35. doi: 10.1016/j.eururo.2009.01.004. Epub 2009 Jan 13. PMID 19150582
- [Background] Brossner C, Pycha A, Toth A, Mian C, Kuber W. Does extended lymphadenectomy increase the morbidity of radical cystectomy? BJU Int. 2004 Jan;93(1):64-6. doi: 10.1111/j.1464-410x.2004.04557.x. PMID 14678370
- [Background] Perera M, McGrath S, Sengupta S, Crozier J, Bolton D, Lawrentschuk N. Pelvic lymph node dissection during radical cystectomy for muscle-invasive bladder cancer. Nat Rev Urol. 2018 Nov;15(11):686-692. doi: 10.1038/s41585-018-0066-1. PMID 30104615
- [Background] Gschwend JE, Heck MM, Lehmann J, Rubben H, Albers P, Wolff JM, Frohneberg D, de Geeter P, Heidenreich A, Kalble T, Stockle M, Schnoller T, Stenzl A, Muller M, Truss M, Roth S, Liehr UB, Leissner J, Bregenzer T, Retz M. Extended Versus Limited Lymph Node Dissection in Bladder Cancer Patients Undergoing Radical Cystectomy: Survival Results from a Prospective, Randomized Trial. Eur Urol. 2019 Apr;75(4):604-611. doi: 10.1016/j.eururo.2018.09.047. Epub 2018 Oct 15. PMID 30337060
- [Background] Froehner M, Novotny V, Heberling U, Rutsch L, Litz RJ, Hubler M, Koch R, Baretton GB, Wirth MP. Relationship of the number of removed lymph nodes to bladder cancer and competing mortality after radical cystectomy. Eur Urol. 2014 Dec;66(6):987-90. doi: 10.1016/j.eururo.2014.07.046. Epub 2014 Aug 19. PMID 25150172
- [Background] Jeong IG, You D, Kim JW, Song C, Hong JH, Ahn H, Kim CS. Outcomes of single lymph node positive urothelial carcinoma after radical cystectomy. J Urol. 2011 Jun;185(6):2085-90. doi: 10.1016/j.juro.2011.02.056. Epub 2011 Apr 15. PMID 21496833
- [Background] Lenis AT, Lec PM, Michel J, Brisbane W, Golla V, Sharma V, Gollapudi K, Blumberg J, Chamie K. Predictors of adequate lymph node dissection in patients with non-muscle invasive bladder cancer undergoing radical cystectomy and effect on survival. Urol Oncol. 2020 Oct;38(10):796.e7-796.e14. doi: 10.1016/j.urolonc.2020.04.027. Epub 2020 May 20. PMID 32446641
- [Background] Abdollah F, Sun M, Schmitges J, Djahangirian O, Tian Z, Jeldres C, Perrotte P, Shariat SF, Montorsi F, Karakiewicz PI. Stage-specific impact of pelvic lymph node dissection on survival in patients with non-metastatic bladder cancer treated with radical cystectomy. BJU Int. 2012 Apr;109(8):1147-54. doi: 10.1111/j.1464-410X.2011.10482.x. Epub 2011 Aug 24. PMID 21883849
- [Background] Bruins HM, Skinner EC, Dorin RP, Ahmadi H, Djaladat H, Miranda G, Cai J, Daneshmand S. Incidence and location of lymph node metastases in patients undergoing radical cystectomy for clinical non-muscle invasive bladder cancer: results from a prospective lymph node mapping study. Urol Oncol. 2014 Jan;32(1):24.e13-9. doi: 10.1016/j.urolonc.2012.08.015. Epub 2013 Feb 6. PMID 23395238
- [Background] Papalia R, Simone G, Grasso R, Augelli R, Faiella E, Guaglianone S, Cazzato R, Del Vescovo R, Ferriero M, Zobel B, Gallucci M. Diffusion-weighted magnetic resonance imaging in patients selected for radical cystectomy: detection rate of pelvic lymph node metastases. BJU Int. 2012 Apr;109(7):1031-6. doi: 10.1111/j.1464-410X.2011.10446.x. Epub 2011 Aug 25. PMID 21883835
- [Background] Li Y, Diao F, Shi S, Li K, Zhu W, Wu S, Lin T. Computed tomography and magnetic resonance imaging evaluation of pelvic lymph node metastasis in bladder cancer. Chin J Cancer. 2018 Jan 26;37(1):3. doi: 10.1186/s40880-018-0269-0. PMID 29370848
- [Background] Del Giudice F, Barchetti G, De Berardinis E, Pecoraro M, Salvo V, Simone G, Sciarra A, Leonardo C, Gallucci M, Catalano C, Catto JWF, Panebianco V. Prospective Assessment of Vesical Imaging Reporting and Data System (VI-RADS) and Its Clinical Impact on the Management of High-risk Non-muscle-invasive Bladder Cancer Patients Candidate for Repeated Transurethral Resection. Eur Urol. 2020 Jan;77(1):101-109. doi: 10.1016/j.eururo.2019.09.029. Epub 2019 Nov 5. PMID 31699526
- [Background] Fragkoulis C, Glykas I, Papadopoulos G, Ntoumas K. Multiparametric MRI in differentiation between muscle invasive and non-muscle invasive urinary bladder cancer with vesical imaging reporting and data system (VI-RADS) application. Br J Radiol. 2020 May 1;93(1109):20200025. doi: 10.1259/bjr.20200025. Epub 2020 Mar 11. No abstract available. PMID 32160006
- [Background] Ueno Y, Takeuchi M, Tamada T, Sofue K, Takahashi S, Kamishima Y, Hinata N, Harada K, Fujisawa M, Murakami T. Diagnostic Accuracy and Interobserver Agreement for the Vesical Imaging-Reporting and Data System for Muscle-invasive Bladder Cancer: A Multireader Validation Study. Eur Urol. 2019 Jul;76(1):54-56. doi: 10.1016/j.eururo.2019.03.012. Epub 2019 Mar 26. PMID 30922688
- [Background] Giacalone NJ, Shipley WU, Clayman RH, Niemierko A, Drumm M, Heney NM, Michaelson MD, Lee RJ, Saylor PJ, Wszolek MF, Feldman AS, Dahl DM, Zietman AL, Efstathiou JA. Long-term Outcomes After Bladder-preserving Tri-modality Therapy for Patients with Muscle-invasive Bladder Cancer: An Updated Analysis of the Massachusetts General Hospital Experience. Eur Urol. 2017 Jun;71(6):952-960. doi: 10.1016/j.eururo.2016.12.020. Epub 2017 Jan 9. PMID 28081860
- [Background] Garcia-Perdomo HA, Montes-Cardona CE, Guacheta M, Castillo DF, Reis LO. Muscle-invasive bladder cancer organ-preserving therapy: systematic review and meta-analysis. World J Urol. 2018 Dec;36(12):1997-2008. doi: 10.1007/s00345-018-2384-6. Epub 2018 Jun 25. PMID 29943218
- [Background] Kulkarni GS, Hermanns T, Wei Y, Bhindi B, Satkunasivam R, Athanasopoulos P, Bostrom PJ, Kuk C, Li K, Templeton AJ, Sridhar SS, van der Kwast TH, Chung P, Bristow RG, Milosevic M, Warde P, Fleshner NE, Jewett MAS, Bashir S, Zlotta AR. Propensity Score Analysis of Radical Cystectomy Versus Bladder-Sparing Trimodal Therapy in the Setting of a Multidisciplinary Bladder Cancer Clinic. J Clin Oncol. 2017 Jul 10;35(20):2299-2305. doi: 10.1200/JCO.2016.69.2327. Epub 2017 Apr 14. PMID 28410011
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542